CLINICAL TRIAL: NCT00346450
Title: Autologous ex Vivo Conjunctival Epithelial Cell Expansion for Ocular Surface
Brief Title: Autologous ex Vivo Conjunctival Epithelial Cell Expansion for Ocular Surface Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: International Stem Cell Forum (Other); National Medical Research Council (NMRC), Singapore (Other Government); Singapore Eye Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R198/24/2000
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Pterygium; Ocular Surface Disease; Stevens Johnson Syndrome; Chemical Injury
Keywords: Culture; Conjunctiva; transplantation; pterygium; ocular surface
MeSH Terms: conditions — Pterygium; Stevens-Johnson Syndrome

INTERVENTIONS:
Procedure: Cultivated conjunctival transplantation

SUMMARY:
To evaluate the use of cultivated conjunctival epithelial equivalents for the treatment of ocular diseases

DETAILED DESCRIPTION:
Ex-vivo autologous conjunctiva expansion on human amniotic membrane (HAM), followed by clinical transplantation surgery

Preparation of HAM. Human amniotic membrane (HAM) prepared for human use will be obtained from the Singapore Eye Bank. HAM will be rapidly thawed in a 37oC water bath, and washed with phosphate buffered saline. The amniotic epithelium will be removed using a combination of Dispase digestion and mechanical scraping. Complete removal of the amniotic epithelial cells will be confirmed by microscopy. The HAM is then placed on a culture plate, with the basement-membrane side up, and incubated with DMEM at 37oC in an atmosphere of 5% CO2 and 95% air overnight before use.

Ex-vivo expansion of conjunctival cells on HAM. A forniceal conjunctival biopsy will be performed in patients undergoing pterygium surgery. The tissue will be cultured on the HAM either as a cell suspension or as explants, with the methods described above. The media is changed every 2 days and the culture is maintained for 2-3 weeks. The cells will form a confluent sheet and begin to stratify and differentiate. The tissue will then be raised to an air-liquid interface to promote differentiation.

Histological analysis. The conjunctival epithelial cell sheets on the amniotic membrane will be examined by light microscopy. Samples of the tissue will be fixed and processed with the use of standard histological procedures and stained with H&E and PAS reagents. Electron microscopic examination will be carried for the tissue. The sections will also be subjected to immunohistochemical analysis for cytokeratin markers.

Clinical Transplantation of cultivated conjunctival epithelial cells on HAM

Preparation of cultivated conjunctival cells on amniotic membrane Patients with various ocular surface disorders will be selected for the initial series of transplantations. All patients will undergo full counselling for informed consent for the procedures. A forniceal conjunctival biopsy will be performed on the contralateral healthy eye. PI will perform the transplantations of autologous conjunctival sheet grown on human amniotic membrane in these patients. The diseased area will be excised using the standard surgical technique. The defect will be covered with the sheet of cultured conjunctival cells on the HAM with the epithelial side up. The graft is secured to the adjacent conjunctiva with interrupted 8/0 vicryl sutures. A planotherapeutic bandage contact lens is placed to protect the tissue from lid trauma. Topical steroid and antibiotic eyedrops will be administered daily to reduce the ocular inflammation. Survival of conjunctiva on the amniotic membrane will be closely monitored and patients will be followed-up at 3 monthly intervals up to one year. During these visits, these patients will have anterior segment photographs taken and fluorescein staining to monitor the progress of healing.

Transplantations may also be carried out on selected patients with ocular surface disease, for example, ocular cicatricial pemphigoid, Stevens Johnson syndrome and alkali injury. For these severe conditions, this procedure may prove to be an important adjunct to other procedures, such as limbal stem cell transplantation. If the initial study is successful, a randomised clinical trial comparing this procedure with conventional conjunctival autografting and conventional amniotic membrane transplantation will be planned. Therefore if found to be successful, transplantation of cultured conjunctival cells on HAM may eventually be used as a primary procedure or as an adjunctive procedure for these visually debilitating conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ocular surface disorders, e.g. primary pterygium, scheduled for elective surgical excision
2. Indications for surgery will be the presence of ocular surface symptoms in the affected eye, loss of visual acuity from visual axis obscuration or irregular astigmatism, or cosmesis.
3. Only one eye of a patient will be eligible for study entry.
4. Patients who are adult males and females who are aged 21 or older, and are considered mentally sound
5. Patients who are willing to undergo long-term follow-up, as outlined in this protocol
6. Patients who have signed an informed consent form that has been approved by the SNEC Ethics Committee.

Exclusion Criteria:

1. Patients less than 21 years of age
2. Patients who are incapable, either by law or of mental state, of giving consent in their own right
3. Patients who are either unable or unwilling to keep scheduled appointments and adhere to the other aspects of the protocol
4. Patients who are pregnant or breastfeeding
5. Patients with a history of drug allergy
6. Patients who have received an investigational drug within 28 days preceding surgery
7. Patients with intraocular pressure over 21 mmHg or history of ocular hypertension or glaucoma
8. Patients who are documented to be steroid responders

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2001-10; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Epithelialisation
Graft integrity
Resolution of inflammation
Visual acuity
Complications

SECONDARY OUTCOMES:
Degree of scarring

CONTACTS AND LOCATIONS:
Overall Officials: Leonard P Ang, FRCS, Principal Investigator — SNEC, NUS; Donald T Tan, FRCS, Principal Investigator — SNEC, SERI, NUS
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Result] Ang LP, Tan DT, Beuerman RW, Lavker RM. Development of a conjunctival epithelial equivalent with improved proliferative properties using a multistep serum-free culture system. Invest Ophthalmol Vis Sci. 2004 Jun;45(6):1789-95. doi: 10.1167/iovs.03-1361. PMID 15161841
- [Result] Ang LP, Tan DT, Phan TT, Li J, Beuerman R, Lavker RM. The in vitro and in vivo proliferative capacity of serum-free cultivated human conjunctival epithelial cells. Curr Eye Res. 2004 May;28(5):307-17. doi: 10.1076/ceyr.28.5.307.28677. PMID 15287367